CLINICAL TRIAL: NCT05240729
Title: Ultrasound Guided Retroclavicular Approach Versus Costoclavicular Approach of Infraclavicular Brachial Plexus Block for Upper Limb Surgeries
Brief Title: Using Ultrasound in Infraclavicular in Upper Limb Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Rowayda Nabil gaber, MD, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 53:2021
Record Dates: First submitted 2022-02-06; First posted 2022-02-15 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Upper Limb Surgeries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Retroclavicular (Active Comparator): Retroclavicular approach to the infraclavicular region, the probe will be placed below and perpendicular to the clavicle, in a paramedian sagittal plane, medial to the coracoid process, to obtain a short-axis view of the cords of the brachial plexus and the axillary vessels. The needle will then be inserted in the supraclavicular fossa, approximately 1 cm posteriorly to the clavicle, and advanced in plane and strictly parallel to the ultrasound transducer. After passing the initial blind zone of about 2 cm caused by the acoustic shadow of the clavicle, the needle tip will be constantly seen, until it will be positioned posterior to the axillary artery.
  Interventions: Procedure: Infraclavicular brachial plexus block
- Costoclavicular (Active Comparator): A new approach to the infraclavicular block The ultrasound transducer will be placed parallel and inferior to the clavicle and angled cephalad to optimize the ultrasound view. The block needle will be inserted in-plane from a lateral to medial direction into the costoclavicular space and the entire drug will be deposited in this location
  Interventions: Procedure: Infraclavicular brachial plexus block
- Classic (Active Comparator): Infraclavicular brachial plexus block (ICPB) ultrasound probe will be placed near the lower edge of the clavicle, and a transverse view of the subclavian artery and vein will be visualized. Using a needle guide, the needle will be advanced under real-time ultrasound guidance, and local anaesthetic will be injected near the subclavian artery, 15 mm medially and 15 mm laterally to the artery. The extent of sensory and motor block will be evaluated at 30 minutes after the injection
  Interventions: Procedure: Infraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Infraclavicular brachial plexus block — Using ultrasound in 3different techniques of infraclavicular brachial plexus block

SUMMARY:
Comparison of 3 approach of infraclavicular brachial plexus

DETAILED DESCRIPTION:
Comparison of retroclavicular & costoclavicular and classic type of infraclavicular brachial plexus block for upper limb surgeries

ELIGIBILITY:
Inclusion Criteria:

* age: between 18 and 60 years ASA I and II BMI between 18 and 35 surgeries to forearm and hand

Exclusion Criteria:

* patient refusal pregnancy allergy to local anaesthetics local infection neuropathy ,coagulopathy anatomical abnormality in clavicular region

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Motor and sensory block success rate | 30 min
  Success rate 30 min after local anasthetic injections

CONTACTS AND LOCATIONS:
Overall Officials: Jozef zekry, MD, Study Chair — Minia University
Locations (1):
- Facutly of Medicine, Minya, Egypt